CLINICAL TRIAL: NCT03099694
Title: Noninvasive Ventilation for Preterm Neonates With Respiratory Distress Syndrome: a Multi-center Randomized Controlled Trial
Brief Title: NHFOV vs. NCPAP as a Primary Treatment to Neonatal Respiratory Distress Syndrome(NRDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xingwang Zhu (Other)
Collaborators: Guiyang Maternity and Child Health Care Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Children's Hospital of Chongqing Medical University (Other); Chongqing Maternal and Child Health Hospital (Other); The Second Hospital of Shandong University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Hunan Children's Hospital (Other Government); Zhengzhou Children's Hospital, China (Other); Chengdu Women's and Children's Central Hospital (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); Kunming Children's Hospital (Other); Chongqing Three Gorges Central Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); University of Southern California (Other); Vilnius University (Other); Children's Hospital of Fudan University (Other); Guangdong Women and Children Hospital (Other); Nanjing Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xingwang Zhu, Director of neonatology, Jiulongpo No.1 People's Hospital
Organization: Jiulongpo No.1 People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jiulongpo People's Hospital
Record Dates: First submitted 2016-11-17; First posted 2017-04-04 (Actual); Results first posted 2019-06-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Preterm Infants
Keywords: NRDS; nHFOV; nCPAP; preterm infants
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nCPAP (Active Comparator): nasal continuous positive airway pressure (nCPAP) - as a primary mode of ventilation in premature infants with RDS
  Interventions: Procedure: nasal continuous positive airway pressure (nCPAP)
- nHFOV (Experimental): noninvasive high-frequency ventilation (nHFOV) as a primary mode of ventilation in premature infants with RDS
  Interventions: Procedure: noninvasive high-frequency ventilation (nHFOV)

INTERVENTIONS:
Procedure: noninvasive high-frequency ventilation (nHFOV) — NHFOV will be provided by a high frequency ventilator (CNO, Medin, Germany or SLE 5000, UK). NHFOV will be provided via binasal prongs.
  Arms: nHFOV
Procedure: nasal continuous positive airway pressure (nCPAP) — Infants assigned to the NCPAP group will be started on a pressure of 6 cmH2O (range: 6-8 cmH2O) by CPAP system (CNO Medin, Germany, Carefusion, USA)
  Arms: nCPAP

SUMMARY:
The investigators compared advantages and disadvantages of two forms of noninvasive respiratory support -noninvasive high-frequency oscillatory ventilation (nHFOV) or nasal continuous positive airway pressure (nCPAP) -as a primary mode of ventilation in premature infants with RDS．

DETAILED DESCRIPTION:
Background: Invasive mechanical ventilation is associated with development of adverse pulmonary and non-pulmonary outcomes in very low birth weight infants. Various modes of non-invasive respiratory support are being increasingly used to minimize the incidence of bronchopulmonary dysplasia (BPD). The aim of this trials to compare the effect of noninvasive high-frequency oscillatory ventilation (NHFOV) and nasal continuous positive airway pressure (NCPAP) in preterm infants with respiratory distress syndrome (RDS) as a primary noninvasive ventilation support mode.

Methods/Design:In this multicenter, randomized, controlled trial, 300 preterm infants at gestational age (GA) less than 34 weeks with a diagnosis of RDS will be randomized to NHFOV or NCPAP as a primary mode of non-invasive respiratory support. Study will be conducted in 18 tertiary neonatal intensive care units in China.

The primary outcome is the need for invasive mechanical ventilation (IMV)during the first 7 days after enrollment in preterm infants randomized to the two groups. The secondary outcomes include days of hospitalization, days on noninvasive respiratory support, days on IMV, days on supplemental oxygen, mortality, need for surfactant, incidence of retinopathy of prematurity(ROP) and bronchopulmonary dysplasia(BPD), occurrence of abdominal distention, air leaks, intraventricular hemorrhage (IVH ≥ grade 3) and necrotizing enterocolitis (NEC> II stage). Other secondary outcomes include scores of Bayley Scales of Infant Development at 2 months and 2 years of corrected age.

ELIGIBILITY:
Inclusion criteria:

(1)Gestational age (GA) is from 26 to 34 weeks; (2) diagnosis of RDS. The diagnosis of RDS will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and chest X-ray findings; (3) RDS Silverman score>5; (4) informed parental consent has been obtained.

Exclusion criteria

(1) severe RDS requiring early intubation according to the American Academy of Pediatrics guidelines for neonatal resuscitation7; (2)major congenital malformations or complex congenital heart disease; (3) group B hemolytic streptococcus pneumonia, septicemia, pneumothorax, pulmonary hemorrhage; (4) cardiopulmonary arrest needing prolonged resuscitation; (5) transferred out of the NICUs without treatment.

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD, Study Director — Third Military Medical University
Locations (1):
- Xingwang Zhu, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Dr. Kris Sekar, Professor of Pediatrics, Oklahoma University Medical Center, Oklahoma, Dr. Jatinder Bhatia, Professor of Pediatrics, Medical College of Georgia, Georgia Health Sciences University, Augusta, Georgia, and Dr. Rowena Cayabyab, MD., MPH (Biostatistics and Epidemiology) Assistant Professor of Pediatrics, Keck School of Medicine of the University of Southern California, Los Angeles, California will serve as DSMB members. Dr. Cayabyab will also serve as consultant for statistical analysis.

REFERENCES:
- [Derived] Zhu X, Feng Z, Liu C, Shi L, Shi Y, Ramanathan R; NHFOV study group. Nasal High-Frequency Oscillatory Ventilation in Preterm Infants with Moderate Respiratory Distress Syndrome: A Multicenter Randomized Clinical Trial. Neonatology. 2021;118(3):325-331. doi: 10.1159/000515226. Epub 2021 Apr 7. PMID 33827081
- [Derived] Zhu XW, Shi Y, Shi LP, Liu L, Xue J, Ramanathan R; NHFOV Study Group. Non-invasive high-frequency oscillatory ventilation versus nasal continuous positive airway pressure in preterm infants with respiratory distress syndrome: Study protocol for a multi-center prospective randomized controlled trial. Trials. 2018 Jun 14;19(1):319. doi: 10.1186/s13063-018-2673-9. PMID 29898763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May, 2017, through July, 2018, a total of 18 centers screened 2509 infants, of which 1385 were eligible. We recruited 340 infants (170 in each group), to account for dropouts. Finally, 302 infants completed the trial (152 in NHFOV; 150 in NCPAP group.)
Pre-assignment Details: 1045 Did not undergo randomization
  * 663 Refused to participate
  * 382 NHFOV devices not available
Groups:
- nCPAP: infants receive primary non-invasive respiratory support by mean of nCPAP
- nHFOV: infants receive primary non-invasive respiratory support by mean of NHFOV
Period: Overall Study
Arm/Group | nCPAP | nHFOV
Started | 170 | 170
Completed | 150 | 152
Not Completed | 20 | 18
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Lost to Follow-up | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- nHFOV: infants receive primary non-invasive respiratory support by mean of NIPPV
- Total: Total of all reporting groups
Arm/Group | nCPAP | nHFOV | Total
Number analyzed (Participants) | 150 | 152 | 302
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 30.9 (1.8) | 30.6 (1.7) | 30.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 61 | 132
  Male | 79 | 91 | 170
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Multiple birth [Count of Participants; unit: Participants] — Mothers of infants
  Participants | 57 | 36 | 93
Antenatal steroids [Count of Participants; unit: Participants] — Mothers of infants
  Participants | 101 | 105 | 206
Cesarean delivery [Count of Participants; unit: Participants] — Mothers of infants
  Participants | 81 | 89 | 170
Premature rupture of membranes>18h [Count of Participants; unit: Participants] — Mothers of infants
  Participants | 61 | 59 | 120
Gestational diabetes mellitus [Count of Participants; unit: Participants] — Mothers of infants
  Participants | 10 | 10 | 20
Birth Weight [Mean (Standard Deviation); unit: g] | 1582 (343) | 1564 (367) | 1572 (351)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required Intubation
Description: The criteria for endotracheal mechanical ventilation were as follows: severe respiratory acidosis (PaCO2 > 60 mmHg with pH<7.20), severe apnea and bradycardia (defined as recurrent apnea with > 3 episodes per hour associated with heart rate < 100/min, a single episode of apnea that required bag and mask ventilation), hypoxia (FiO2>0.5 with PaO2<50mmHg), severe respiratory distress, neonatal pulmonary hemorrhage, and cardiopulmonary arrest without effective resuscitation needing continued ventilation and rescue
Time Frame: during the first 7 days after birth
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 26 | 15

2. Secondary Outcome: the Incidence of Intraventricular Hemorrhage (IVH, ≥ Grade Ⅲ)
Description: The criteria for intraventricular hemorrhage (IVH, ≥ grade Ⅲ): intraventricular hemorrhage with ventricular dilatation and intraventricular hemorrhage with paren- ehymal hemorrhage. Intraventricular hemorrhage (≥ grade Ⅲ) is worse outcome.
Time Frame: first two months after birth
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 2 | 4

3. Secondary Outcome: the Incidence of Pneumothorax
Description: the incidence of pneumothorax
Time Frame: during non-invasive ventilation, up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 1 | 3

4. Secondary Outcome: the Incidence of Neonatal Necrotizing Enterocolitis(>Stage II)
Description: The criteria for neonatal necrotizing enterocolitis(>stage II): Unequivocal malfunction of the gastrointestinal tract is demonstrated clinically and by radiographic evaluation. Other disorders such as malrotation and volvulus and Hirschsprung's disease must be excluded.
  Neonatal necrotizing enterocolitis(>stage II) is worse outcome
Time Frame: during non-invasive ventilation, up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 7 | 11

5. Secondary Outcome: the Incidence of Retinopathy of Prematurity (>Stage II)
Description: The criteria for Retinopathy of prematurity (>Stage II); extraretinal fibrovascular proliferation neovascularization extends from ridge into the vitreous. Retinopathy of prematurity (>Stage II) is worse outcome.
Time Frame: at a post-menstrual age of 36 weeks or at discharge
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 9 | 7

6. Secondary Outcome: The Score of Bayley Scales of Infant Development
Description: scores of Bayley Scales of Infant Development at 2 months old and 2 years old
Time Frame: 30 months
Reporting Status: Not Posted, anticipated posting 2021-09

7. Secondary Outcome: the Incidence of Bronchopulmonary Dysplasia(BPD)
Description: BPD was defined according to the National Institutes of Health consensus definition: Need for O2 supplementation(FiO2>0.21) for at least 28 days after birth.
  BPD is worse outcome.
Time Frame: at a post-menstrual age of 36 weeks or at discharge
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 15 | 17

8. Secondary Outcome: the Incidence of Abdominal Distention
Description: Abdominal circumference increase 2 centimeter during non-invasive ventilation
Time Frame: during non-invasive ventilation, up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 19 | 26

9. Secondary Outcome: The Time of Non-invasive Ventilation
Description: Hours
Time Frame: during non-invasive ventilation, up to 30 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
hours | 81.0 [40.0 to 166.0] | 78.5 [48.0 to 163.5]

10. Secondary Outcome: Length of Hospitalization
Description: Days
Time Frame: during hospitalization, up to 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
days | 29.0 [19.0 to 41.0] | 31.0 [18.5 to 41.0]

11. Secondary Outcome: Predischarge Mortality
Time Frame: during hospitalization, up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 4 | 6

12. Secondary Outcome: Length of O2 Therapy
Description: Days
Time Frame: during hospitalization, up to 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
days | 7.0 [4.0 to 17.0] | 8.0 [4.0 to 17.0]

13. Secondary Outcome: Number of Participants With Thick Secretions Causing an Airway Obstruction
Description: determined by the clinician
Time Frame: during non-invasive ventilation, up to 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP | nHFOV
Number analyzed (Participants) | 150 | 152
Participants | 8 | 21

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | nHFOV | nCPAP
All-Cause Mortality (participants affected / at risk) | 6/152 | 4/150
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150
Other Adverse Events (participants affected / at risk) | 0/152 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03099694/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03099694/ICF_001.pdf